CLINICAL TRIAL: NCT04190823
Title: A Phase I Study to Evaluate the Safety,Tolerability and Pharmacokinetics of RC98 For Injection in Subjects With Advanced Malignant Solid Tumors
Brief Title: A Study of RC98 in Subjects With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC98-C001
Record Dates: First submitted 2019-12-01; First posted 2019-12-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC98 (Experimental)
  Interventions: Drug: RC98

INTERVENTIONS:
Drug: RC98 — Participants will be allocated to one of the following dose groups: 0.003, 0.03, 0.3, 2.5, 5.0, 10.0, 15.0 and 20.0 mg/kg, and receive one treatment of RC98 followed by 28 days of dose limited toxicity (DLT) observation period.
  Other Names: RC98 for Injection

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of RC98 for injeciton in subjects with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Diagnosed with histologically or cytologically-confirmed locally advanced or metastatic solid tumors.
* Measurable lesion according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment:

Cardiac ejection fraction ≥ 50 %. Hemoglobin ≥ 90g/L; Absolute neutrophil count ≥ 1.5×10^9 /L Platelets ≥ 100×10^9 /L; Total bilirubin ≤ 1.5× ULN and ≤ 1.5× ULN with hepatic metastasis; AST and ALT ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN; INR, APTT and PT ≤ 1.5× ULN; TSH or FT4 or FT3 in (1±10%) ULN.

* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Known hypersensitivity to the components of RC98 for injection.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia).
* Pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* History of receiving any research drug treatment within 4 weeks prior to trial treatment.
* History of major surgery, chemotherapy or radiotherapy within 4 weeks of planned start of trial treatment.
* History of arterial / venous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism, occurred within 6 months before study medication.
* NYHA Class III heart failure.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Currently known active infection with HIV or tuberculosis.
* Diagnosed with HBsAg , HBcAb positive and HBV DNA copy positive, or HCVAb positive.
* Uncontrolled hypertension, diabetes, pulmonary fibrosis, acute lung disease, interstitial lung disease, or cirrhosis;
* Treated with corticosteroids or other immunosuppressants for the autoimmune disease within 14 days prior to the study treatment.
* Existing active, or have experienced autoimmune diseases that may recur (eg: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis Disease, etc.) or subjects with these disease risks.
* Pregnancy or lactation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial.
* Presence of primary tumors of the nervous system, brain metastases and / or cancerous meningitis.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* History of receiving immune-enhancing therapy (eg, alpha-interferon, interleukin-2), hormone therapy, traditional Chinese medicine treatment, or palliative radiotherapy for bone metastases within 2 weeks of planned start of trial treatment.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | From the day of ICF sign to 28 days after the day of the last treatment
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v4.03
Maximum Tolerated dose of RC98 | 12 months
  The dose level in which >= 2 out of 6 patients have dose-limiting toxicity (DLT). The MTD is defined as the previous dose level.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 15 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Progression Free Survival (PFS) | 15 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No